CLINICAL TRIAL: NCT04597086
Title: The Effects of Bright White Light Therapy on Fatigue, Sleep, Distress, Depression and Anxiety in the Hospitalized Leukemia Patient
Brief Title: Bright White Light Therapy for the Improvement of Sleep, Fatigue, Distress, Depression, and Anxiety in Hospitalized Leukemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Shelly Brown, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-20091; NCI-2020-07234 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Acute Leukemia; Recurrent Leukemia; Refractory Leukemia
MeSH Terms: conditions — Leukemia | interventions — Practice Guidelines as Topic; Standard of Care; Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (BWLT, best practice) (Experimental): Patients receive BWLT over 30 minutes in addition to standard of care daily during hospital stay.
  Interventions: Other: Best Practice; Procedure: Bright White Light Therapy; Other: Survey Administration
- Group II (standard of care) (Active Comparator): Patients receive standard of care during hospital stay.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Procedure: Bright White Light Therapy — Receive BWLT
  Arms: Group I (BWLT, best practice)
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial investigates how well bright white light therapy works in improving sleep, fatigue, distress, depression, and anxiety, side effects that are often experienced during an intense leukemia treatment regimen, in hospitalized leukemia patients. Bright white light therapy may help to control these symptoms, and information from this study may help doctors and nurses learn more about methods for decreasing these symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy of bright white light therapy (BWLT) on fatigue in patients diagnosed with leukemia during their hospitalization.

SECONDARY OBJECTIVES:

I. To assess the efficacy of BWLT on sleep disturbance in patients diagnosed with leukemia during their hospitalization.

I. To assess the efficacy of BWLT on anxiety in patients diagnosed with leukemia during their hospitalization.

III. To assess the efficacy of BWLT on depression in patients diagnosed with leukemia during their hospitalization.

IV. To assess the efficacy of BWLT on distress in patients diagnosed with leukemia during their hospitalization.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive BWLT over 30 minutes in addition to standard of care daily during hospital stay.

GROUP II: Patients receive standard of care during hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Acute Leukemia Unit for an anticipated stay of 3 weeks or longer
* English speaking
* Able to comprehend and sign a consent form
* Able to read and complete surveys
* Alert and oriented
* Without BWLT for seven days prior to initiating the trial

Exclusion Criteria:

* Current eye disorders which is defined as:

  * Iritis, uveitis, keratitis, cataract, glaucoma, macular degeneration, retinal detachment, or retinitis pigmentosa
* Diagnosed bipolar disorder
* Persons with pacemakers

  * The manufacturer of the BWLT unit used for this study mentions the light unit contains magnets

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Level of fatigue | Up to one month after discharge
  Will be assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue. Will fit a mixed model of fatigue as a function of time and group.

SECONDARY OUTCOMES:
Sleep disturbance | Up to one month after discharge
  Will be assessed by PROMIS-Sleep Disturbance. Will fit a mixed model.
Anxiety | Up to one month after discharge
  Will be assessed by General Anxiety Disorder-7. Will fit a mixed model.
Depression | Up to one month after discharge
  Will be assessed by Patient Health Questionnaire Depression Scale. Will fit a mixed model.
Distress | Up to one month after discharge
  Will be assessed by Distress Thermometer. Will fit a mixed model.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Brown, MS, APRN-CNS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT04597086/ICF_000.pdf